CLINICAL TRIAL: NCT05769907
Title: Motivational to Weight Loss Version 1 (MWL v.1): Protocol for a Feasibility Single-arm, Open-label Clinical Trial of a Motivational Interviewing, Stages and Processes of Change-based Intervention for Weight Loss in Adults
Brief Title: Protocol for a Feasibility of a Motivational Interviewing for Weight Loss in Adults
Acronym: MWL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Adriane Ribeiro Rosa, Professor, Hospital de Clinicas de Porto Alegre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20220209; 59573622300005327 (Other: CAAE)
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Obesity
Keywords: Obesity; Transtheoretical Model; P-Weight; S-Weight; Change talk; Motivational interviewing
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Study setting The study was carried on by the Laboratory of Molecular Psychiatry at Hospital Clinic of Porto Alegre (HCPA), Brazil. The study will consist of face-to-face sessions performed in the Clinical Research Center (CPC) of the HCPA and online sessions performed through the platform Teams.
  This project complies with the guidelines presented in SPIRIT 2013 "Standard protocol items: Recommendations for Interventional Trials," an international protocol that aims to improve the completeness of studies, producing recommendations for a minimum set of items to be addressed. The 2013 SPIRIT Statement includes a 33-item checklist .
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): The single-arm pilot study will be a feasibility study of the Motivation to Lose Weight version 1 (MLW v.1). The study includes presential and online sessions. Participants will be recruited through advertisements on social media and selected according to the inclusion criteria. Participants will receive 8 sessions of approximately 30-45 minutes of motivational interviewing (MI) according to the processes of change in weight loss, as measured by the S-Weight scale.
  Interventions: Behavioral: Intervention Group

INTERVENTIONS:
Behavioral: Intervention Group — The study will consist of one session per week for 8 weeks, during which the participant will receive MI for 30-45 minutes. All participants will receive the MI intervention according to their readiness to lose weight measured by means the P-weight and S-weight at the beginning of each session.

SUMMARY:
Abstract Introduction: This pilot study will determine the recruitment feasibility, retention, and adhesion for a motivational interviewing program for weight loss in adults according to the processes of change in weight loss.

Methods and Analysis: The single-arm pilot study will be a feasibility study of the Motivation to Lose Weight version 1 (MLW v.1). The study includes presential and online sessions. Participants will be recruited through advertisements on social media and selected according to the inclusion criteria. Participants will receive 8 sessions of approximately 30-45 minutes of motivational interviewing (MI) according to the processes of change in weight loss, as measured by the S-Weight scale. The results will be evaluated at the beginning and the end of the program, which will last 8 weeks. The primary outcome of the study is feasibility. The intervention will be feasible if adherence to the proposed activities in the sessions is greater than 70%, we can recruit 10 patients within 8 weeks, the proportion of interested people and registered participants is greater than 30%, and more than 75% of participants attend the final study visit. The secondary outcome is weight loss, fat mass percentage, muscle mass, waist and hip measurements, and the scores of behavioral scales.

Ethics and discussion: The feasibility of this project consists of proposing an individualized intervention based on MI strategy(s) for each participant, according to the stage of readiness, and thus, help to evolve in the process of losing weight. This intervention aims to increase the participant's confidence level to implement actions that lead to the progression of behavior and, consequently, the action and maintenance of the lost weight. This study was approved by the Research Ethics Committee (REC) of the Hospital de Clínicas de Porto Alegre (HCPA) under number 20220209 CAAE 59573622300005327.

DETAILED DESCRIPTION:
The study will consist of one session per week for 8 weeks, during which the participant will receive MI for 30-45 minutes. All participants will receive the MI intervention according to their readiness to lose weight measured by means the P-weight and S-weight at the beginning of each session.

In session one, sociodemographic and clinical information will be collected through a structured interview as well clinical assessment including the following scales: the stage of change to lose weight (S-Weight), symptoms of depression (PROMIS depression v. 8.1a, ), anxiety (PROMIS anxiety v.8.1a, ), psychosocial functioning (FAST ), binge eating (TCAP ), current food intake (24-hours food recall, ), and cognitive process used while losing weight (P-Weight ). In addition, the first session will collect information regarding the participant's body weight, body fat, free fat mass, and waist and hip circumference.

As participants will be in the precontemplation or contemplation stage of change at the beginning of the study, the goals of the first session will be: a) develop participant rapport; b) develop the discrepancy, that is, understand the distance between what the participant wants to change and the actions are taken; c) roll with resistance, that is, do not conflict during the dialogue; d) avoid the correction reflex, that is, avoid correcting something the interviewee says, even if it is technically incorrect or not plausible; e) valuing and validating the person, that is, emphasizing points in the participant's speech to increase their self-confidence; f) establish an agenda of issues to be deal with that are related to being overweight or obese. All these objectives remain in subsequent sessions. To accomplish those goals, the interviewer will use the MI process called "explore," which leads to the topic the participant wants to discuss. The interviewer will use strategies such as open questions, affirmations, reflections, abstracts, exploring discrepancies, informing with permission, explore values and objectives based on the participants' speech in order to elicit from the person their different motives for the desired change . Each session will be registered following the Session Registration Form .

From sessions two to seven, the sessions will take place online through the platform Teams, and the participant will answer the S-weight scale to identify the actual stage of change to lose weight at the beginning of each session. In case of the participant is in the precontemplation, contemplation or preparation phases, the goals in the session will be a) encourage the participant to talk about the reasons that favor him to change and not to change; b) focus on the positive motives to change; c) Increase the participants' confidence, that is, explain that the style of this approach takes into account their autonomy, and thus, any and all decision-making will be shared and not directed from the interviewer to he/she, also because a basic premise of MI is that people are experts on themselves; d) extract from the participant how he/she could make the change, anticipating what it would be like if he/she had already made the change; e) show options for the participant to choose from, based on their own answers; f) stimulate through questions and reflections that the participant himself talks about his/her abilities, this increases the confidence that he is capable of doing things; g) prepare the participant for the action phase; h) predict difficulties; and i) prevent relapse. However, if the participant is in the action, maintenance, or relapse phase, the goals will be to a) stimulate the participant to develop solutions to promote autonomy and confidence in the decision-making process; b) reinforce the commitment to change; c) recall the participants' values through reflections; d) validate the actions already taken, even if they are damage reductions; e) support self-confidence; f) increase support network; g) prevent relapse; and h) consolidate the gains from the changes made.

The goals established in sessions two to seven will be pursued by the interviewer by using the MI process "focus," "evoke," and "plan". Focus will direct the conversation toward the possibility of change, creating a discrepancy between the participants' current actions and their broader life goals and values . Evoking will stimulate the participant to talk about their motivations for change. Planning includes helping the participant to identify a goal, building an action plan, and anticipating difficulties. The interviewer will use strategies such as closed questions, open questions, reflection, importance rule, and trust ruler.

In the last session, the participant will attend an in-person session for the measurement of body weight, body fat, free fat mass, waist, and hip circumference, as well as the assessment of the same clinical scales used in the first session). In addition, the participant will fill in a questionnaire regarding the interviewer's attitude during the sessions, which will indicate the compliance of the researcher with the MI approach.

ELIGIBILITY:
Inclusion Criteria:

Aged 18-60; BMI from 25-34.90 (Kg/m²); Residents of Porto Alegre and nearby regions; No weight loss treatment in the last 6 months; Pre-contemplation or contemplation phase for changing body weight when responding to the S-Weight scale; Stable body weight in the last 3 months (<2% loss); Access to Teams platform; Have access to a body weight scale.

Exclusion Criteria:

Major surgery in the last 3 months; Diagnosed eating disorder; Use of mood stabilizer drugs or antipsychotics, antiobesity or adjuvants in weight control, as well as corticoids (prednisone and similar) in doses greater than 10 mg per day; Dietary treatment for weight loss in the last 6 months; Myocardial infarction or angioplasty in the last 3 months, with chronic kidney disease or undergoing dialysis; with chronic liver failure (Ascites), with congestive heart failure, undergoing treatment for cancer or with the Human Immunodeficiency Virus (HIV); Pregnant and lactating women.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — people over 18 and under 60
Enrollment: 54 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is to test the feasibility and acceptability of the pilot study | 8 weeks
  Adherence rate, Recruitment rate, Retention rates

SECONDARY OUTCOMES:
percentage of weight loss body | 8 weeks
  5% of baseline
number of participants who progressed through stages of change in weight loss | 8 weeks
  70% of participants progress through the change stage

CONTACTS AND LOCATIONS:
Overall Officials: Quênia de Carvalho, Author, Principal Investigator — HC Porto Alegre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burgess E, Hassmen P, Welvaert M, Pumpa KL. Behavioural treatment strategies improve adherence to lifestyle intervention programmes in adults with obesity: a systematic review and meta-analysis. Clin Obes. 2017 Apr;7(2):105-114. doi: 10.1111/cob.12180. Epub 2017 Feb 15. PMID 28199047
- [Background] de Freitas PP, de Menezes MC, Dos Santos LC, Pimenta AM, Ferreira AVM, Lopes ACS. The transtheoretical model is an effective weight management intervention: a randomized controlled trial. BMC Public Health. 2020 May 11;20(1):652. doi: 10.1186/s12889-020-08796-1. PMID 32393214
- [Background] Di Noia J, Prochaska JO. Dietary stages of change and decisional balance: a meta-analytic review. Am J Health Behav. 2010 Sep-Oct;34(5):618-32. doi: 10.5993/ajhb.34.5.11. PMID 20524891
- [Background] Hayotte M, Negre V, Gray L, Sadoul JL, d'Arripe-Longueville F. The transtheoretical model (TTM) to gain insight into young women's long-term physical activity after bariatric surgery: a qualitative study. Obes Surg. 2020 Feb;30(2):595-602. doi: 10.1007/s11695-019-04220-9. PMID 31654341
- [Background] Karintrakul S, Angkatavanich J. A randomized controlled trial of an individualized nutrition counseling program matched with a transtheoretical model for overweight and obese females in Thailand. Nutr Res Pract. 2017 Aug;11(4):319-326. doi: 10.4162/nrp.2017.11.4.319. Epub 2017 Jun 22. PMID 28765778
- [Background] Tanikawa Y, Kimachi M, Ishikawa M, Hisada T, Fukuhara S, Yamamoto Y. Association between work schedules and motivation for lifestyle change in workers with overweight or obesity: a cross-sectional study in Japan. BMJ Open. 2020 Apr 30;10(4):e033000. doi: 10.1136/bmjopen-2019-033000. PMID 32354776
- [Background] Hardcastle SJ, Taylor AH, Bailey MP, Harley RA, Hagger MS. Effectiveness of a motivational interviewing intervention on weight loss, physical activity and cardiovascular disease risk factors: a randomised controlled trial with a 12-month post-intervention follow-up. Int J Behav Nutr Phys Act. 2013 Mar 28;10:40. doi: 10.1186/1479-5868-10-40. PMID 23537492
- [Background] Ismail K, Stahl D, Bayley A, Twist K, Stewart K, Ridge K, Britneff E, Ashworth M, de Zoysa N, Rundle J, Cook D, Whincup P, Treasure J, McCrone P, Greenough A, Winkley K. Enhanced motivational interviewing for reducing weight and increasing physical activity in adults with high cardiovascular risk: the MOVE IT three-arm RCT. Health Technol Assess. 2019 Dec;23(69):1-144. doi: 10.3310/hta23690. PMID 31858966
- [Background] Moss EL, Tobin LN, Campbell TS, von Ranson KM. Behavioral weight-loss treatment plus motivational interviewing versus attention control: lessons learned from a randomized controlled trial. Trials. 2017 Jul 25;18(1):351. doi: 10.1186/s13063-017-2094-1. PMID 28743313
- [Background] Suire KB, Kavookjian J, Feiss R, Wadsworth DD. Motivational Interviewing for Weight Management Among Women: a Meta-Analysis and Systematic Review of RCTs. Int J Behav Med. 2021 Aug;28(4):403-416. doi: 10.1007/s12529-020-09934-0. Epub 2020 Oct 20. PMID 33083891
- [Background] Makin H, Chisholm A, Fallon V, Goodwin L. Use of motivational interviewing in behavioural interventions among adults with obesity: A systematic review and meta-analysis. Clin Obes. 2021 Aug;11(4):e12457. doi: 10.1111/cob.12457. Epub 2021 May 6. PMID 33955152
- [Background] Toral N, Slater B. [Transtheoretical model approach in eating behavior]. Cien Saude Colet. 2007 Nov-Dec;12(6):1641-50. doi: 10.1590/s1413-81232007000600025. Portuguese. PMID 18813500
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Andres A, Saldana C, Gomez-Benito J. Establishing the stages and processes of change for weight loss by consensus of experts. Obesity (Silver Spring). 2009 Sep;17(9):1717-23. doi: 10.1038/oby.2009.100. Epub 2009 Apr 9. PMID 19360014
- [Background] Duran Aguero S, Araneda J, Ahumada D, Silva Rojas J, Bonacich RB, Caichac A, Salamanca MF, Villarroel P, Fernandez E, Pacheco V, Martinovic PA, Wilson W, Neira AM, Encina C, Tilleria JM. A Multicenter Study Evaluating the Stages of Change in Food Consumption with Warning Labels among Chilean University Students. Biomed Res Int. 2020 Jan 16;2020:2317929. doi: 10.1155/2020/2317929. eCollection 2020. PMID 32461968
- [Background] Andres A, Saldana C, Beeken RJ. Assessment of processes of change for weight management in a UK sample. Obes Facts. 2015;8(1):43-53. doi: 10.1159/000373900. Epub 2015 Jan 29. PMID 25765163
- [Background] Rosa AR, Andreazza AC, Sanchez-Moreno J, Gazalle FK, Santin A, Stein A, Barros HM, Vieta E, Kapczinski F. Validation of the Portuguese version of the Lithium Attitudes Questionnaire (LAQ) in bipolar patients treated with lithium: cross-over study. Clin Pract Epidemiol Ment Health. 2006 Nov 22;2:32. doi: 10.1186/1745-0179-2-32. PMID 17121674
- [Background] Andres A, Saldana C, Gomez-Benito J. The transtheoretical model in weight management: validation of the processes of change questionnaire. Obes Facts. 2011;4(6):433-42. doi: 10.1159/000335135. Epub 2011 Nov 25. PMID 22248993
- [Background] de Castro NFC, de Melo Costa Pinto R, da Silva Mendonca TM, da Silva CHM. Psychometric validation of PROMIS(R) Anxiety and Depression Item Banks for the Brazilian population. Qual Life Res. 2020 Jan;29(1):201-211. doi: 10.1007/s11136-019-02319-1. Epub 2019 Oct 9. PMID 31598816
- [Background] Rosa AR, Sanchez-Moreno J, Martinez-Aran A, Salamero M, Torrent C, Reinares M, Comes M, Colom F, Van Riel W, Ayuso-Mateos JL, Kapczinski F, Vieta E. Validity and reliability of the Functioning Assessment Short Test (FAST) in bipolar disorder. Clin Pract Epidemiol Ment Health. 2007 Jun 7;3:5. doi: 10.1186/1745-0179-3-5. PMID 17555558
- [Background] Resnicow K, McMaster F. Motivational Interviewing: moving from why to how with autonomy support. Int J Behav Nutr Phys Act. 2012 Mar 2;9:19. doi: 10.1186/1479-5868-9-19. PMID 22385702
- [Background] Forsberg L, Kallmen H, Hermansson U, Berman AH, Helgason AR. Coding counsellor behaviour in motivational interviewing sessions: inter-rater reliability for the Swedish Motivational Interviewing Treatment Integrity Code (MITI). Cogn Behav Ther. 2007;36(3):162-9. doi: 10.1080/16506070701339887. PMID 17852172
- [Background] Brug J, Spikmans F, Aartsen C, Breedveld B, Bes R, Fereira I. Training dietitians in basic motivational interviewing skills results in changes in their counseling style and in lower saturated fat intakes in their patients. J Nutr Educ Behav. 2007 Jan-Feb;39(1):8-12. doi: 10.1016/j.jneb.2006.08.010. PMID 17276321
- [Background] Ziebart C, MacDermid J, Bryant D, Szekeres M, Suh N. Hands-Up program: protocol for a feasibility randomised controlled trial of a combined 6-week exercise and education intervention in adults aged 50-65 with a distal radius fracture. BMJ Open. 2021 Jul 30;11(7):e046122. doi: 10.1136/bmjopen-2020-046122. PMID 34330854
- [Background] Browne RH. On the use of a pilot sample for sample size determination. Stat Med. 1995 Sep 15;14(17):1933-40. doi: 10.1002/sim.4780141709. PMID 8532986
- [Background] Hertzog MA. Considerations in determining sample size for pilot studies. Res Nurs Health. 2008 Apr;31(2):180-91. doi: 10.1002/nur.20247. PMID 18183564
- [Background] Teare MD, Dimairo M, Shephard N, Hayman A, Whitehead A, Walters SJ. Sample size requirements to estimate key design parameters from external pilot randomised controlled trials: a simulation study. Trials. 2014 Jul 3;15:264. doi: 10.1186/1745-6215-15-264. PMID 24993581
- [Background] Nymberg P, Ekvall Hansson E, Stenman E, Calling S, Sundquist K, Sundquist J, Zoller B. Pilot study on increased adherence to physical activity on prescription (PAP) through mindfulness: study protocol. Trials. 2018 Oct 17;19(1):563. doi: 10.1186/s13063-018-2932-9. PMID 30333052
- [Background] Carels RA, Darby L, Cacciapaglia HM, Konrad K, Coit C, Harper J, Kaplar ME, Young K, Baylen CA, Versland A. Using motivational interviewing as a supplement to obesity treatment: a stepped-care approach. Health Psychol. 2007 May;26(3):369-74. doi: 10.1037/0278-6133.26.3.369. PMID 17500624
- [Background] Woo S, Park KH. Motivating Children and Adolescents in Obesity Treatment. J Obes Metab Syndr. 2020 Dec 30;29(4):260-269. doi: 10.7570/jomes20026. PMID 32843587
- [Background] Erol S, Erdogan S. Application of a stage based motivational interviewing approach to adolescent smoking cessation: the Transtheoretical Model-based study. Patient Educ Couns. 2008 Jul;72(1):42-8. doi: 10.1016/j.pec.2008.01.011. Epub 2008 Mar 4. PMID 18304775
- [Background] Miller WR, Rollnick S. Ten things that motivational interviewing is not. Behav Cogn Psychother. 2009 Mar;37(2):129-40. doi: 10.1017/S1352465809005128. PMID 19364414
- [Background] Wilson GT, Schlam TR. The transtheoretical model and motivational interviewing in the treatment of eating and weight disorders. Clin Psychol Rev. 2004 Jul;24(3):361-78. doi: 10.1016/j.cpr.2004.03.003. PMID 15245836
- [Background] Maula A, Kendrick D, Kai J, Griffiths F. Evidence generated from a realist synthesis of trials on educational weight loss interventions in type 2 diabetes mellitus. Diabet Med. 2021 Jan;38(1):e14394. doi: 10.1111/dme.14394. Epub 2020 Oct 8. PMID 32871624
- [Background] Culliford A, Bradbury J. A cross-sectional survey of the readiness of consumers to adopt an environmentally sustainable diet. Nutr J. 2020 Dec 9;19(1):138. doi: 10.1186/s12937-020-00644-7. PMID 33298065
- [Background] Clark PG, Greene GW, Blissmer BJ, Lees FD, Riebe DA, Stamm KE. Trajectories of Maintenance and Resilience in Healthful Eating and Exercise Behaviors in Older Adults. J Aging Health. 2019 Jun;31(5):861-882. doi: 10.1177/0898264317746264. Epub 2017 Dec 12. PMID 29254440
- [Result] Chopra S, Malhotra A, Ranjan P, Vikram NK, Sarkar S, Siddhu A, Kumari A, Kaloiya GS, Kumar A. Predictors of successful weight loss outcomes amongst individuals with obesity undergoing lifestyle interventions: A systematic review. Obes Rev. 2021 Mar;22(3):e13148. doi: 10.1111/obr.13148. Epub 2020 Nov 16. PMID 33200547
- [Result] Lecube A, Sanchez E, Andres A, Saldana C, Morales MJ, Calanas A, Minambres I, Pellitero S, Cordido F, Bueno M, Caixas A, Vilarrasa N; Obesity Group of the Spanish Society of Endocrinology and Nutrition (GOSEEN). Assessing Motivational Stages and Processes of Change for Weight Management Around Bariatric Surgery: a Multicenter Study. Obes Surg. 2019 Oct;29(10):3348-3356. doi: 10.1007/s11695-019-04001-4. PMID 31209830
- [Result] Armstrong MJ, Mottershead TA, Ronksley PE, Sigal RJ, Campbell TS, Hemmelgarn BR. Motivational interviewing to improve weight loss in overweight and/or obese patients: a systematic review and meta-analysis of randomized controlled trials. Obes Rev. 2011 Sep;12(9):709-23. doi: 10.1111/j.1467-789X.2011.00892.x. Epub 2011 Jun 21. PMID 21692966
- [Result] Durrer Schutz D, Busetto L, Dicker D, Farpour-Lambert N, Pryke R, Toplak H, Widmer D, Yumuk V, Schutz Y. European Practical and Patient-Centred Guidelines for Adult Obesity Management in Primary Care. Obes Facts. 2019;12(1):40-66. doi: 10.1159/000496183. Epub 2019 Jan 23. PMID 30673677
- [Result] Knight KM, McGowan L, Dickens C, Bundy C. A systematic review of motivational interviewing in physical health care settings. Br J Health Psychol. 2006 May;11(Pt 2):319-32. doi: 10.1348/135910705X52516. PMID 16643702
- [Result] Ceccarini M, Borrello M, Pietrabissa G, Manzoni GM, Castelnuovo G. Assessing motivation and readiness to change for weight management and control: an in-depth evaluation of three sets of instruments. Front Psychol. 2015 May 11;6:511. doi: 10.3389/fpsyg.2015.00511. eCollection 2015. PMID 26029126
- [Result] Mastellos N, Gunn LH, Felix LM, Car J, Majeed A. Transtheoretical model stages of change for dietary and physical exercise modification in weight loss management for overweight and obese adults. Cochrane Database Syst Rev. 2014 Feb 5;2014(2):CD008066. doi: 10.1002/14651858.CD008066.pub3. PMID 24500864
- [Result] Prochaska JO, DiClemente CC, Norcross JC. In search of how people change. Applications to addictive behaviors. Am Psychol. 1992 Sep;47(9):1102-14. doi: 10.1037//0003-066x.47.9.1102. PMID 1329589
- See also: PSS Health: Power and Sample Size for Health Researchers [Internet]. [cited 11 de fevereiro de 2021] — https://hcpa-unidade-bioestatistica.shinyapps.io/PSS_Health